CLINICAL TRIAL: NCT01325558
Title: A Phase I, Open-Label, Multi-center, Competitive Enrollment and Dose-escalation Study of ALT-836 in Combination With Gemcitabine for Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of ALT-836 in Combination With Gemcitabine for Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altor BioScience (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-836-02-10
Record Dates: First submitted 2011-03-09; First posted 2011-03-30 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Locally Advanced Malignant Neoplasm; Malignant Solid Tumour
Keywords: cancer; tissue factor; solid tumor; ovarian cancer; breast cancer; non-small cell lung cancer; colon cancer; pancreatic cancer; head and neck cancer; prostate cancer; soft-tissue sarcoma; metastatic; gemcitabine; anti-tumor; venous thromboembolism
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Pancreatic Neoplasms; Head and Neck Neoplasms; Prostatic Neoplasms; Sarcoma; Neoplasm Metastasis; Venous Thromboembolism | interventions — ALT-836; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: ALT-836 in combination with gemcitabine — Study participants will receive up to four courses of a 28-day biochemotherapy with the study drug (ALT-836) and gemcitabine. Each treatment course consists of five doses of ALT-836 (on Day 1, 4, 8, 15 and 22) and three doses of gemcitabine (Day 1, 8 and 15). Participants with persistent responses will receive additional two cycles, three doses each, of standard of care gemcitabine therapy.

SUMMARY:
This is a Phase I, open-label, multi-center, competitive enrollment and dose-escalation study of ALT-836 in combination with standard of care gemcitabine in participants who have locally advanced or metastatic solid tumors. The purpose of this study is to determine the maximum tolerated dose (MTD), and to assess the safety and pharmacokinetic profile of ALT-836 given with gemcitabine. The clinical benefit, progression-free survival and overall survival of study participants will also be assessed.

DETAILED DESCRIPTION:
Tissue Factor (TF) is over-expressed in most cancer types. Results from many recent studies have suggested a key role for TF in the development of cancer-associated thrombosis, tumor growth, tumor angiogenesis, and tumor metastasis. ALT-836, a recombinant human-chimeric monoclonal antibody, is designed as a direct TF antagonist to block TF displayed by cancers and to inhibit cancer-associated venous thromboembolism, tumor growth, tumor angiogenesis and tumor metastasis. In numerous pre-clinical studies in laboratory animals, including non-human primates, ALT-836 exhibits potent anti-tumor, anti-thrombotic and anti-inflammatory activities with a remarkable safety profile. In humans, ALT-836, administered as a single bolus and monotherapy in patients with coronary artery disease (CAD) and acute lung injury/acute respiratory distress syndrome (ALI/ARDS), is safe and exhibits anti-coagulant and anti-inflammatory effects. A Phase II study using a multi-dose regimen of ALT-836 is being conducted in patients with ALI/ARDS. In the dose-escalation study described in this protocol, the investigators will assess the safety and determine the maximum tolerated dose (MTD) of ALT-836 in combination with gemcitabine in patients with advanced malignancies known to overexpress TF and in which venous thromboembolism is a major complication.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed
* Locally advanced or metastatic non-hematologic malignancies
* Measureable
* Refractory to standard therapies or single agent gemcitabine is indicated as a standard treatment option

PRIOR/CONCURRENT THERAPY:

* No concurrent radiotherapy, chemotherapy, immunotherapy or other investigational agents
* Must have recovered from side effects of prior therapies

PATIENT CHARACTERISTICS:

Life expectancy

* > 12 weeks

Performance Status

* ECOG 0 or 1

Bone Marrow Reserve

* Absolute Neutrophil count (AGC/ANC) ≥ 1,500/uL
* Platelets ≥ 100,000/uL
* Hemoglobin > 9 g/dL

Renal Function

* Calculated Glomerular filtration rate (GFR) > 59mL/min/1.73M^2

Hepatic Function

* Total bilirubin ≤ 1.5 X ULN
* AST, ALT, and ALP ≤ 3 X ULN or ≤ 5.0 x ULN, if liver metastasis exists
* PT INR ≤ 1.5 X ULN

Cardiovascular

* No history of clinically significant vascular disease
* No New York Heart Association (NYHA) Class > II heart failure

Hematologic

* No history of bleeding disorders
* No evidence of bleeding diathesis or coagulopathy
* No presence of clinically significant hemoptysis or hematuria, presence of serious non-healing wound or ulceration, or signs of other bleeding
* No evidence of a tumor invasion of any major blood vessel
* No trauma with increased risk of life-threatening bleeding or history of severe head trauma or intracranial surgery within two months of study entry

Surgery/Procedures

* No major surgery or open biopsy within 28 days before drug infusion or evidence of active bleeding postoperatively
* No plan for any major surgery during treatment period
* No presence or requirement of an epidural catheter or lumbar puncture within 48 hours prior to each dose of study treatment
* No anticipation of receiving an epidural catheter or a lumbar puncture within 48 hours after each dose of study treatment

Excluded Medications or Treatment Regimens

* Unfractionated heparin of > 15,000 units/day within 8 hours prior to each dose of study treatment
* Low-molecular weight heparin at a higher dose than recommended for prophylactic used or required within 20 hours prior to each dose of study treatment
* Warfarin used or required within 48 hours prior to each dose of study treatment and the prothrombin time (INR) exceeded the upper limit of normal range
* Direct thrombin inhibitors or Xa inhibitors
* Acetylsalicylic acid used or required within 72 hours prior to each dose of study treatment
* Clopidogrel bisulfate used or required within 48 hours prior to each dose of study treatment
* Anticipated requirement for anti-platelet or anti-coagulant agents excluding non-aspirin NSAID within 48 hours following study treatment infusion

Other

* No active systemic infection requiring parenteral antibiotic therapy
* No history of or presence of a CNS disease
* No history of allergic reactions to compounds of similar chemical or biologic composition
* Not HIV positive
* No women who are pregnant or nursing
* A negative serum pregnancy test if female
* Patients, both females and males, with reproductive potential must agree to use effective contraceptive measures for the duration of the study
* No history of significant renal, endocrinologic, metabolic, immunologic or hepatic disease
* No evidence of psychiatric illness/social situations
* Other illness that in the opinion of the investigator would exclude the patient from participating
* Must provide informed consent and HIPAA authorization and comply with protocol-specified procedures and follow-up evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ALT-836 in combination with gemcitabine | 18 months
Safety Profile | 18 months
  Number and severity of treatment related AEs that occur or worsen after the first dose of study treatment
Clinical Benefit | 18 months
  Number of participants with complete response, partial response or stable disease
Progression Free Survival | 36 months
  Number of participants with 9-month, 12-month, 18-month, 24-month, 30-month or 36-month progression-free survival

SECONDARY OUTCOMES:
Overall Survival | 36 months
  Number of participants with 9-month, 12-month, 18-month, 24-month, 30-month or 36-month overall survival
Pharmacokinetics | 18 months
  Area under the plasma concentration-time curve from time zero to infinity (AUC) and the half-life of ALT-836

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Rochester Medical Center, James P. Wilmot Cancer Center, Rochester, New York
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No